CLINICAL TRIAL: NCT06251934
Title: Real-World Patient Characteristics, Treatment Patterns, and Clinical Outcomes Among Patients With BRAF-Positive Metastatic Melanoma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS66
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: BRAF-positive Metastatic Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- Patients with high tumor burden (HTB)
- Patients with low tumor burden (LTB)
- Patients with central nervous system (CNS) metastases
- Patients with without CNS metastases
- 1L IO-refractory patients

SUMMARY:
This was a retrospective, longitudinal, observational study conducted using the Flatiron Health electronic health record (EHR)-derived database. BRAF+ advanced or metastatic (i.e., stage III or IV) melanoma patients treated at oncology practices across the US were identified for potential inclusion. All included patients were aged ≥18 years and required to have a diagnosis of melanoma (International Classification of Diseases (ICD)-9 172.x & ICD-10 C43 or D03x), a pathologic unresectable stage III or IV diagnosis, subsequent first-line (1L) treatment with either immunotherapy (IO) (nivolumab, pembrolizumab, ipilimumab + nivolumab) or targeted therapy (TT) dafratenib + trametinib (dab/tram) on or after 01 January 2014, and evidence of a BRAF-positive result at any point in time.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of melanoma (ICD-9 172x & ICD-10 C43 or D03x)
* ≥2 documented clinical encounters on different days in the Flatiron network on or after 01 January 2011
* Pathologic unresectable stage III or IV at initial diagnosis after 01 January 2011, or earlier stage disease accompanied by development of a first locoregional recurrence after 01 January 2011
* Diagnosis of MM after 01 January 2011
* Evidence of a BRAF-positive result at any point in time
* Treatment with one of the following 1L therapies on or after 01 January 2014:

  * IO (nivolumab, pembrolizumab, or ipilimumab + nivolumab)
  * TT (dab/tram)
* At least 18 years of age at the time of initiation of 1L therapy
* At least 6-months of continuous follow-up from the time of initiation of 1L therapy

Exclusion Criteria:

* Lacking relevant unstructured documents (i.e., information such as free text from a physician note or pathology report that is captured systematically during the data abstraction process) in the Flatiron Health database
* Evidence of non-skin melanoma (ocular, subungual, mucosal, palmar, plantar)
* Documented receipt of a clinical study drug, defined as any uncancelled order, administration, or oral episode for a clinical study drug for cancer at any time prior to or during 1L treatment
* Presence of leptomeningeal disease (ICD-9 198.4 & ICD-10 C79.32 or C79.49)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 785 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Mean age of 1L dab/tram-treated BRAF+ MM patients | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients who identify per sex | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients per race category | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients per ethnicity category | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients per geographic region | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients per type of medical practice | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients per insurance type | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients with an Eastern Cooperative Oncology Group (ECOG) score of 0, 1, 2, 3, or 4 | Baseline
  ECOG performance status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scores can range from a lower value of 0 (fully active, able to carry on all pre-disease performance without restriction) up to 5 (dead).
Number and percentage of 1L dab/tram-treated BRAF+ MM patients per location of metastatic site | Baseline
Alanine aminotransferase (ALT) levels in 1L dab/tram-treated BRAF+ MM patients | Baseline
Aspartate aminotransferase (AST) levels in 1L dab/tram-treated BRAF+ MM patients | Baseline
Lactate dehydrogenase (LDH) levels in 1L dab/tram-treated BRAF+ MM patients | Baseline
Number and percentage of 1L dab/tram-treated BRAF+ MM patients treated with 2L therapy | Up to approximately 2 years
Time from the start of 1L dab/tram therapy until the start of 2L therapy | Up to approximately 2 years
Real-world progression-free survival (rwPFS) for 1L dab/tram-treated BRAF+ MM patients | Up to approximately 2 years
  rwPFS was defined as the time from the start of 1L dab/tram therapy until first progression or death from any cause.
Overall survival (OS) for 1L dab/tram-treated BRAF+ MM patients | Up to approximately 2 years
  OS was defined as the time from the start of 1L dab/tram therapy until death from any cause.

SECONDARY OUTCOMES:
Mean age of 1L IO-refractory patients with BRAF+ MM | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM who identify per sex | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM per race category | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM per ethnicity category | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM per geographic region | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM per type of medical practice | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM per insurance type | Baseline
Number and percentage of 1L IO-refractory patients with BRAF+ MM with an ECOG score of 0, 1, 2, 3, or 4 | Baseline
  ECOG performance status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). Scores can range from a lower value of 0 (fully active, able to carry on all pre-disease performance without restriction) up to 5 (dead).
Number and percentage of 1L IO-refractory patients with BRAF+ MM per location of metastatic site | Baseline
Alanine aminotransferase (ALT) levels in 1L IO-refractory patients with BRAF+ MM | Baseline
Aspartate aminotransferase (AST) levels in 1L IO-refractory patients with BRAF+ MM | Baseline
Lactate dehydrogenase (LDH) levels in 1L IO-refractory patients with BRAF+ MM | Baseline
Time from the first disease progression until next disease progression in 1L IO-refractory patients with BRAF+ MM | Up to approximately 2 years
Number and proportion of patients remaining on 1L IO therapy following disease progression | Up to approximately 2 years
Time patients remained on 1L IO therapy following disease progression | Up to approximately 2 years
Number and percentage of patients treated with 2L therapy, overall and by therapy type | Up to approximately 2 years
Time from the start of 1L IO until the start of 2L therapy | Up to approximately 2 years
Time from the first disease progression until the start of 2L therapy | Up to approximately 2 years
rwPFS for 1L IO-refractory patients with BRAF+ MM | Up to approximately 2 years
  rwPFS was defined as the time from the first disease progression until next progression or death from any cause.
OS for 1L IO-refractory patients with BRAF+ MM | Up to approximately 2 years
  OS was defined as the time from the first disease progression until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States